CLINICAL TRIAL: NCT05468671
Title: Department of Anesthesiology, Cancer Hospital of the University of Chinese Academy of Sciences（Zhejiang Cancer Hospital), Research Center for Neuro-Oncology Interaction , Institute of Basic Medicine and Cancer, Chinese Academy of Sciences
Brief Title: Clinical Application Value of Remazolam Combined With Sugammadex Sodium in Anesthesia for Endotracheal Surgery Under Bronchoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xie Kangjie, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2020-406
Record Dates: First submitted 2022-07-13; First posted 2022-07-21 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Endobronchial Metastases; Bronchoesophageal Fistula; General Anesthetic Drug Adverse Reaction
MeSH Terms: interventions — remimazolam; Propofol; Rocuronium; Remifentanil; Oxycodone; Sugammadex; Flumazenil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remazolam general anesthesia group (R group) (Experimental): Remazolam 0.4 mg/kg, oxycodone 0.2 mg/kg and rocuronium 0.9 mg/kg were given for anesthesia induction.Group R was given remazolam 1mg/kg/h and remifentanil 6-8ug/kg/h for maintenance.
  Interventions: Drug: Remimazolam; Drug: Rocuronium; Drug: Remifentanil; Drug: oxycodone; Drug: Sugammadex Sodium; Drug: Flumazenil
- Propofol general anesthesia control group (P group) (Active Comparator): Propofol 1.5mg/kg, oxycodone 0.2mg/kg and rocuronium 0.9mg/kg were given for induction of anesthesia.Group P was given propofol 4-8 mg/kg/h and remifentanil 6-8ug/kg/h for anesthesia maintenance.
  Interventions: Drug: Propofol; Drug: Rocuronium; Drug: Remifentanil; Drug: oxycodone; Drug: Sugammadex Sodium

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is a new drug innovation in anesthesia. It combines the properties of two unique drugs already established in anesthesia - Midazolam and remifentanil. It acts on GABA receptors like midazolam and has organ-independent metabolism like remifentanil.
  Arms: Remazolam general anesthesia group (R group)
Drug: Propofol — Propofol is used to put you to sleep and keep you asleep during general anesthesia for surgery or other medical procedures.
  Arms: Propofol general anesthesia control group (P group)
Drug: Rocuronium — Rocuronium is a non-depolarizing neuromuscular blocker
Drug: Remifentanil — Remifentanil is an esterase-metabolized opioid
Drug: oxycodone — Oxycodone is an opiate painkiller.
Drug: Sugammadex Sodium — Sugammadex sodium is an organic sodium salt that is the octasodium salt of sugammadex. Used for reversal of neuromuscular blockade induced by rocuronium and vecuronium in adults undergoing surgery
Drug: Flumazenil — Flumazenil is used to reverse the effects of a benzodiazepine
  Arms: Remazolam general anesthesia group (R group)

SUMMARY:
This study is a prospective, randomized, controlled trial. In this study, 30 patients who underwent endotracheal tumor resection under rigid bronchoscope or stent placement for acquired tracheoesophageal fistula were selected as the subjects. The patients were randomly divided into remazolam general anesthesia group (R group) and propofol general anesthesia control group (P group). Remazolam general anesthesia group (R group): Remazolam 0.4 mg/kg, oxycodone 0.2 mg/kg and rocuronium 0.9 mg/kg were given for anesthesia induction. Propofol general anesthesia control group (P group): Propofol 1.5mg/kg, oxycodone 0.2mg/kg and rocuronium 0.9mg/kg were given for induction of anesthesia. After induction, high-frequency jet ventilation was used in both groups, the respiratory rate was 30-60 times/min, the inspiratory-to-breath ratio was 1:2, and the driving pressure was 0.8-1.0 KPa. Group R was given remazolam 1mg/kg/h and remifentanil 6-8ug/kg/h for maintenance. Group P was given propofol 4-8 mg/kg/h and remifentanil 6-8ug/kg/h for anesthesia maintenance. The dosage of propofol or remazolam was adjusted according to BIS and intraoperative hemodynamic changes. Rocuronium bromide 10 mg was added every half hour. Intraoperative application of vasoactive drugs to maintain mean arterial pressure above 60mmHg to avoid perioperative hypotension. Blood oxygen saturation and end-tidal carbon dioxide were monitored to avoid perioperative hypoxemia and hypercapnia, and warm measures were used to maintain the patient's intraoperative body temperature above 36.0°C. After surgery, group R was treated with sugammadex sodium 2-4 mg/kg to antagonize rocuronium bromide, and 0.5 mg of flumazenil was used to antagonize remazolam by intravenous injection; group P was treated with sugammadex 2-4 mg/kg to antagonize rocuronium.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bronchoscopy endotracheal tumor resection or stenting of acquired tracheoesophageal fistula within a limited time
* >18 Years
* ASA Ⅱ-Ⅳ

Exclusion Criteria:

* <18Years
* Refuse to participate
* A history of schizophrenia, epilepsy, Parkinson's disease or myasthenia gravis;
* Severe hepatic dysfunction (Child-Pugh class C)
* Severe renal dysfunction (requiring dialysis)
* Patients with ASA grade Ⅴ and above
* Emergency Surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Recovery time in seconds | postoperative, 2 hours
  Taking the stop of general anesthesia as the starting point for timing, the time for the patient to correctly complete the three commands of nodding, mouth opening and tongue extension is recorded, with seconds as the timing unit

SECONDARY OUTCOMES:
Modified Brice Questionnaire in YES or NO | postoperative，24 hours
  Modified Brice interview over quality assurance techniques in detecting intraoperative awareness.
Intraoperative mean arterial blood pressure in mmHg | Intraoperative，4hours
  Fluctuations in intraoperative systolic, diastolic pressures and mean arterial pressure will be recorded
Perioperative Nutrition Status Assessment Scale (PONS) in YES or NO | Baseline, 1 year
  PONS is a modified version of the malnutrition universal screening tool and determines the presence of nutrition risk based on BMI, recent body weight loss, decrement of dietary intake, and preoperative albumin concentration.
Onset time in seconds | Induction of anesthesia，10 minutes
  The time from the start of peripheral intravenous injection of general anesthetic to the patient's loss of consciousness. Time is measured in seconds.
The incidence of Postoperative delirium in rate | postoperative，24 hours
  The proportion of cases of postoperative delirium in the enrolled patients
Intraoperative heart rate in beats per minute | Intraoperative，4hours
  Fluctuations in intraoperative heart rate will be recorded
The incidence of postoperative vomiting in rate | postoperative，24 hours
  The proportion of cases of postoperative vomiting in the enrolled patients

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hanzhou, China

IPD SHARING:
Plan to Share IPD: No